CLINICAL TRIAL: NCT03396263
Title: Randomized Control Trial to Evaluate the Effectiveness of Online Versus Face-to-face Nutrition Advice in Kuwait (The EatWellQ8 Study)
Brief Title: Online vs. Face-to-face Nutritional Advice in Kuwait (EatWellQ8)
Acronym: EatWellQ8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor Julie A Lovegrove, University of Reading
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13/17b
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Dietary Modification; Dietary Habits
Keywords: Personalised nutrition; Mobile web application
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online personalised advice (Experimental): Online (web-based) delivery of personalised dietary, weight and physical activity advice based on the individual's dietary intake, weight and physical activity levels, generated by the e-Nutri web application. Participants in this group will receive online personalised reports.
  Interventions: Behavioral: Online personalised advice
- Face-to-face personalised advice (Experimental): Face-to-face delivery of personalised dietary, weight and physical activity advice based on the individual's dietary intake, weight and physical activity levels, generated by the e-Nutri web application. Participants in this group will receive nutritional advice face-to-face (in person or via video chat).
  Interventions: Behavioral: Face-to-face personalised advice
- Control (Placebo Comparator): Non-personalised advice Control group. Online (web-based) delivery of non- personalised dietary, weight and physical activity advice based on the UK general health guidelines. This arm will be using the e-Nutri web application. Participants in this group will receive online general recommendations (non- personalised).
  Interventions: Behavioral: Non-personalised advice

INTERVENTIONS:
Behavioral: Non-personalised advice — Provision of online non-personalised advice on dietary intake, weight and physical activity levels. Non-personalised dietary advice for improved food choice based on standard population health guidelines.
  Arms: Control
Behavioral: Online personalised advice — Provision of online personalised advice on dietary intake, weight and physical activity levels. Personalised recommendations for improved food choice based on adherence to an 11-item modified US Alternative Healthy Eating Index (m-AHEI), for weight based on ideal BMI range and for physical activity based on the Baecke questionnaire/results.
  Arms: Online personalised advice
Behavioral: Face-to-face personalised advice — Provision of face-to-face personalised advice on dietary intake, weight and physical activity levels. Personalised recommendations for improved food choice based on adherence to an 11-item modified US Alternative Healthy Eating Index (m-AHEI), for weight based on ideal BMI range and for physical activity based on the Baecke questionnaire/results.
  Arms: Face-to-face personalised advice

SUMMARY:
The EatWellQ8 study aims to investigate the effectiveness of a mobile web application (e-Nutri), capable of delivering automated personalised nutrition advice, compared with face-to-face nutritional advice, in increasing diet quality.

Dietary assessment is via the validated Food4Me FFQ (with an updated user interface that has been designed for better usability) and dietary feedback is derived according to adherence to an 11-item modified US Alternative Healthy Eating Index (m-AHEI).

ELIGIBILITY:
Inclusion Criteria:

* aged > 21 years

Exclusion Criteria:

* aged < 21 years old
* not living in the UK
* pregnant/lactating
* no or limited access to internet
* following a prescribed diet for any reason
* intolerance or food allergy
* subject with diabetes, or any other metabolic disorder or illness that alters nutritional requirements

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2017-12-24 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Dietary change | baseline, 6 weeks, 12 weeks
  Change from baseline in dietary intake at 6 and 12 weeks assessed via a Food Frequency Questionnaire (FFQ). An 11-item modified US Alternative Healthy Eating Index (m-AHEI), which is calculated from the results of the FFQ, will be used to quantify the dietary intake changes.

SECONDARY OUTCOMES:
Weight | baseline, 6 weeks, 12 weeks
  Change from baseline in self-reported weight (kg) at 6 and 12 weeks. Weight variation will be combined with height (constant for adults) and also reported as BMI variation (kg/mˆ2).
Physical activity | baseline, 6 weeks, 12 weeks
  Change from baseline in self-reported physical activity (Baecke questionnaire) at 6 and 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Dasman Diabetes Institute, Kuwait City, Kuwait
- University of Reading, Reading, Berkshire, United Kingdom